CLINICAL TRIAL: NCT01062139
Title: A Randomized, Parallel, Double-blind, Multi-center, Comparative Study to Exploratively Evaluate the Efficacy and Safety of Cosalin® Monotherapy vs. Cosalin® and Xarlin® Combination Therapy in Patients With Allergic Rhinitis
Brief Title: Cosalin® Monotherapy Versus Cosalin® and Xarlin® Combination Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Hyo Hyoung, Lee / CRA, CJ Cheiljedang Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CJ_COS_M01
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — levocetirizine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Petasites extract, levocetirizine (Experimental): Cosalin (Petasites hybridus CO2 extract), Xarlin (levocetirizine) combination therapy group
  Interventions: Drug: Xarlin (Levocetirizine); Drug: Cosalin (Petasites hybridus CO2 extract)
- Cosalin (Petasites hybridus CO2 extract) (Active Comparator): Cosalin monotherapy
  Interventions: Drug: Cosalin (Petasites hybridus CO2 extract)

INTERVENTIONS:
Drug: Xarlin (Levocetirizine) — Combination therapy compared to mono therapy
  Other Names: Cosalin (Petasites hybridus CO2 extract); Xyarin (levocetirizine)
  Arms: Petasites extract, levocetirizine
Drug: Cosalin (Petasites hybridus CO2 extract) — Combination therapy compared to mono therapy

SUMMARY:
Title of Study:

A randomized, parallel, double-blind, multi-center, comparative study to evaluate the efficacy and safety of Cosalin monotherapy versus Cosalin and Xarlin combination therapy in patients with allergic rhinitis

Objective of study:

To exploratively evaluate superiority of combination therapy - twice-daily Cosalin Tab (Petasites hybridus CO2 extract) with once-daily Xarlin Tab (Levocetirizine HCl) - compared to monotherapy of Cosalin with allergic rhinitis subjects.

DETAILED DESCRIPTION:
Number of Subjects:

Total 100 subjects / Each group 50 subjects (combination therapy group, monotherapy group / include 20% of subjects drop out rate)

Test Products:

Cosarlin (Petasites hybridus CO2 extract) 30 mg tablet Xarlin (Levocetirizine HCl) 5 mg tablet

Study Design:

Development Phase: Phase IV Randomized, double blind, active-controlled, multi-center study

The subject, who is to satisfy inclusion criteria and not to satisfy any of exclusion criteria will be allocated 1:1 to combination therapy group or mono therapy group, randomized.

Written informed consent will be obtained from the subjects prior to study entry.

Dose, Mode of administration:

Monotherapy group - Cosalin 30mg tablet two times daily. Combination therapy group - Cosalin 30mg tablet two times daily and Xarlin 5mg tablet once daily.

Duration of Tx:

2 Weeks

Safety Endpoint:

Physical Exam, Adverse Events, Vital Signs at Visit 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female volunteer more than 18 years old and less than 66 years old.
2. A volunteer who is informed about this study and sign the informed consent.
3. A volunteer who is diagnosed perennial allergic rhinitis greater than grade3 at visit 1(screening visit) by allergy skin test or serum IgE antibody assay in 24 months.
4. A volunteer who has score 8 and more than 8 point 4 Total Symptom Score (4TSS - runny nose, nasal congestion, itchy nose, sneezing).

Exclusion Criteria:

1. A volunteer who has hypersensitivity to Levocetirizine or Hydroxyzine
2. A volunteer who has hypersensitivity to Petasites hybridus leaves.
3. A volunteer who has anaphylaxis or hypersensitivity to allergy skin test.
4. A volunteer who has serious renal failure or liver failure. Ingestion of antibiotics during previous two weeks from Visit 1, cause of upper respiratory infection(include paranasal sinus).
5. A volunteer who need to use steroids cause of asthma.
6. A volunteer who is using steroids, decongestants, antihistamine.
7. A volunteer who has rhinitis medicamentosa.
8. A volunteer who has seasonal allergic rhinitis.
9. A volunteer who has Galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption genetic disorder .
10. A volunteer who is an alcoholic or a drug addict.
11. Women who are pregnant, breast-feeding, women who plan to get pregnant during the trial period, or do not use authorized contraceptive methods (e.g: sterilization, intrauterine device, combined use of oral contraceptives and barrier contraceptive, combined use of other hormone delivery systems and barrier contraceptive and combined use of contraceptive cream, jelly or foam and diaphragm or condom) in spite of possibility of pregnancy.
12. A volunteer who has experience to take test products in 1 month.
13. A volunteer who is concluded poor compliance or fail to follow medical instruction

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Compare efficacy improvement of combination therapy group and mono therapy group by percent change of 4 TSS from baseline to end of treatment by investigator. | 2 weeks

SECONDARY OUTCOMES:
Compare percent change of evening reflective 4 TSS from baseline to end of treatment by using patient diary. | 2 weeks
Compare percent change of instantaneous 4 TSS from baseline to end of treatment by using patient diary. | 2 weeks
Compare percent change of evening reflective nasal congestion score from baseline to end of treatment by using patient diary. | 2 weeks
Compare percent change of instantaneous nasal congestion score from baseline to end of treatment by using patient diary. | 2 weeks
Compare percent change of evening reflective 5 TSS (5 TSS - runny nose, itchy nose, sneezing, ocular symptom, nasal congestion)by using patient diary. | 2 weeks
Compare percent change of instantaneous 5 TSS by using patient diary. | 2 weeks
Compare percent change of evening reflective 4 TSS from baseline to each day by using patient diary. | 2 weeks
Compare percent change of instantaneous 4 TSS from baseline to each day by using patient diary. | 2 weeks
Compare improvement of QoL from baseline to end of treatment, by using RQLQ (Rhinoconjunctivitis Quality of Life Questionnaire). | 2 weeks
Compare responder rate (> 50% evening reflective 4TSS improvement) by using patient's diary. | 2 weeks